CLINICAL TRIAL: NCT01443702
Title: Use of Lapis Judaicus to Dissolve Kidney Stones
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pouya Faridi, Principal Investigator, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Shirazums CT-90-5677
Record Dates: First submitted 2011-09-25; First posted 2011-09-30 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Kidney Calculi
Keywords: Kidney Calculi; Iranian traditional medicine; Lapis judaicus
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Lapis judaicus (Active Comparator)
  Interventions: Drug: Lapis Judaicus

INTERVENTIONS:
Drug: Lapis Judaicus — 2 g capsule per day.
  Arms: Lapis judaicus
Drug: Placebo — 2 g capsule per day.
  Arms: Placebo

SUMMARY:
The investigators will investigate the safety and effectiveness of an Iranian traditional medicine regarding its ability to dissolve existing kidney stones. Calcium stone formers will be recruited for a 12 week trial. Each subject will receive Lapis judaicus or placebo in random order. End points are changes in urinary chemistries and stone burden by Ultra sonography / CT scan.

It will be used in proven calcium stone forming adults who are not pregnant. This phase is a double blind, randomized, placebo controlled Entry, first and 12 week 24 hour urine supersaturations, pH and sodium determinations will be collected. Entry and final stone quantification Ultra sonography / CT scan will be performed. End points will be changes in urine chemistry/supersaturation and stone quantitative stone volume.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Mentally competent
* Medically effective birth control if fertile female
* History of calcium containing stone AND current quantifiable stone
* Able to comply with protocol

Exclusion Criteria:

* Prisoner
* Pregnant
* CKD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Stone size after 12 weeks | 8 weeks and 12 weeks
  24 hour urine chemistries 24 hour urine supersaturation Stone quantification CT

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Roozbeh, MD, Study Chair — Shiraz University of Medical Sciences
Locations (1):
- Motahhari Medical Center, Shiraz, Fars, Iran